CLINICAL TRIAL: NCT00550394
Title: Quetiapine Plus Topiramate or Placebo for Bipolar Mania & Alcohol Use in Adolescents & Young Adults
Brief Title: Efficacy and Tolerability of Topiramate in Treatment of Bipolar Mania and Alcohol Use in Adolescents and Young Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Melissa Delbello, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIAAA; R21AA016372 (NIH)
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2014-10

CONDITIONS: Bipolar Disorder; Alcohol Abuse
Keywords: Adolescents
MeSH Terms: conditions — Bipolar Disorder; Alcoholism | interventions — Quetiapine Fumarate; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine and Placebo (Active Comparator): Quetiapine and Placebo
  Interventions: Drug: quetiapine and placebo
- Quetiapine and Topiramate (Experimental): Quetiapine and Topiramate
  Interventions: Drug: Quetiapine and Topiramate

INTERVENTIONS:
Drug: quetiapine and placebo — Dosing Schedule and Titration of Quetiapine: open-label quetiapine beginning day 1 at 100 mg/day titrated to 400 mg/day by the end of week 1
  Dosing Schedule and Titration of Topiramate:
  All subjects will be randomized to topiramate or matching placebo which will be administered in a double-blind manner.
  Topiramate/Placebo titrated from 25 mg twice daily to 150 mg bid by week 4.
  Other Names: Quetiapine
  Arms: Quetiapine and Placebo
Drug: Quetiapine and Topiramate — Dosing Schedule and Titration of Quetiapine:
  open-label quetiapine beginning day 1 at 100 mg/day titrated to 400 mg/day by the end of week 1
  Dosing Schedule and Titration of Topiramate:
  All subjects will be randomized to topiramate or matching placebo which will be administered in a double-blind manner.
  Topiramate/Placebo titrated from 25 mg twice daily to 150 mg bid by week 4.
  Other Names: Topiramate
  Arms: Quetiapine and Topiramate

SUMMARY:
The purpose of this research study is to study the effects (both good and bad) of combining quetiapine and topiramate for treating symptoms of bipolar mania (an illness with periods of elation, excessive excitement, irritability, high energy, racing thoughts, poor sleep, poor judgment, reckless behavior) and to study the effects (both good and bad) of combining quetiapine and topiramate for reducing use of alcohol.

DETAILED DESCRIPTION:
Specific Aim 1: To collect preliminary data regarding the efficacy and tolerability of topiramate for the treatment of alcohol use disorders (alcohol abuse and dependence) in adolescents with bipolar disorder.

Hypothesis 1: We hypothesize that topiramate in combination with quetiapine will lead to greater reduction in alcohol consumption (number of drinks per day, number of drinks per drinking day, and number of heavy drinking days) and greater abstinence (percentage of days abstinent) compared with quetiapine alone.

Specific Aim 2: To obtain preliminary data regarding the efficacy of topiramate for reducing manic symptoms in adolescents with co-occurring alcohol use and bipolar disorders.

Hypothesis 2: We hypothesize that the topiramate in combination with quetiapine will produce greater reduction in Young Mania Rating Scale (YMRS) scores than quetiapine alone.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 12-25 years;
2. DSM-IV-TR83 criteria for bipolar disorder, type I, manic or mixed episode;
3. Young Mania Rating Scale (YMRS)86-88 score of > 16 at screening and baseline visits;
4. DSM-IV-TR83 criteria for current alcohol abuse or dependence;
5. Drinking >8 drinks in 30 days within the previous 6 months while meeting DSM-IV criteria for alcohol abuse or dependence.

   One standard drink is defined as 0.35 liters of beer, 0.15 liters of wine, or 0.04 liters of 80-proof liquor;
6. Fluent in English;
7. Provision of written informed consent/assent; 8) If female and of child bearing potential, agrees to use one of the following method of birth control: complete abstinence, barrier (diaphragm or condom), or oral contraceptive containing > 35 micrograms of ethinyl estradiol (because concomitant use of topiramate and lower estrogen oral contraceptives may lead to contraceptive failure).

Exclusion Criteria:

1. Manic symptoms resulting from acute medical illness or acute intoxication or withdrawal from drugs or alcohol as determined by medical evaluation and rapid symptom resolution;
2. Clinically significant alcohol or drug withdrawal symptoms that have the potential to cause serious consequences as determined by vital signs, the CIWA-Ar,84 and medical evaluation;
3. Any unstable medical illness or laboratory abnormalities > 3 times upper limits of normal;
4. A documented history of mental retardation or an IQ total score < 70 as determined by the Wechsler Abbreviated Scale of Intelligence (WASI),154 administered by a trained psychometrician;
5. Any substance use other than alcohol, nicotine, or cannabis during the 30 days prior to study participation;
6. A positive urine pregnancy test or lactating;
7. History of nephrolithiasis.
8. Treatment with concurrent mood stabilizers, antipsychotics or antidepressants;
9. Treatment with antipsychotics or other mood stabilizers within 72 hours and antidepressants within 5 days prior to randomization;
10. Treatment with fluoxetine within one month;
11. A history of non-response or hypersensitivity to quetiapine or topiramate;
12. Serious suicidal ideation (> 3 on the CDRS-R89 suicide item, or any serious suicide attempt within the prior 60 days as judged by the investigator; 3=has thoughts about suicide or hurting themselves usually when angry);
13. Treatment for substance use during 30 days prior to screening (excluding peer support groups);
14. Court-ordered to substance use treatment;
15. Acute intoxication;
16. History of a medication change during the prior 30 days that may have precipitated manic symptoms;
17. History of a partial response (any improvement) to any existing medications as reported by treating clinician, subjects or legal guardian.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa P DelBello, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 56 study participants were consented for study participation, of which 17 were screen fails.
Pre-assignment Details: 56 study participants were consented for study participation, of which 17 were screen fails.
Groups:
- Quetiapine and Placebo: Quetiapine and Placebo
  quetiapine and placebo: Dosing Schedule and Titration of Quetiapine: open-label quetiapine beginning day 1 at 100 mg/day titrated to 400 mg/day by the end of week 1
  Dosing Schedule and Titration of Topiramate:
  All subjects will be randomized to topiramate or matching placebo which will be administered in a double-blind manner.
  Topiramate/Placebo titrated from 25 mg twice daily to 150 mg bid by week 4.
- Quetiapine and Topiramate: Quetiapine and Topiramate
  Quetiapine and Topiramate: Dosing Schedule and Titration of Quetiapine:
  open-label quetiapine beginning day 1 at 100 mg/day titrated to 400 mg/day by the end of week 1
  Dosing Schedule and Titration of Topiramate:
  All subjects will be randomized to topiramate or matching placebo which will be administered in a double-blind manner.
  Topiramate/Placebo titrated from 25 mg twice daily to 150 mg bid by week 4.
Period: Overall Study
Arm/Group | Quetiapine and Placebo | Quetiapine and Topiramate
Started | 21 | 18
Completed | 9 | 5
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Quitiapine and Placebo: Quetiapine and Placebo
  quetiapine and placebo: Dosing Schedule and Titration of Quetiapine: open-label quetiapine beginning day 1 at 100 mg/day titrated to 400 mg/day by the end of week 1
  Dosing Schedule and Titration of Topiramate:
  All subjects will be randomized to topiramate or matching placebo which will be administered in a double-blind manner.
  Topiramate/Placebo titrated from 25 mg twice daily to 150 mg bid by week 4.
- Quitiapine andTopiramate: Quetiapine and Topiramate
  Quetiapine andTopiramate: Dosing Schedule and Titration of Quetiapine:
  open-label quetiapine beginning day 1 at 100 mg/day titrated to 400 mg/day by the end of week 1
  Dosing Schedule and Titration of Topiramate:
  All subjects will be randomized to topiramate or matching placebo which will be administered in a double-blind manner.
  Topiramate/Placebo titrated from 25 mg twice daily to 150 mg bid by week 4.
- Total: Total of all reporting groups
Arm/Group | Quitiapine and Placebo | Quitiapine andTopiramate | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 18 | 39
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18 (3.1) | 17.7 (2.4) | 17.9 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 24
  Male | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  United States | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Day
Description: Change in self-reported drinks/day (drinks consumed divided by the number of days during that study period).
Time Frame: baseline to 12 weeks or endpoint (up to 11 weeks)
Measure: Mean (Standard Deviation); unit: Drinks per day
Groups:
- Quetiapine + Placebo: Quetiapine + Placebo
  quetiapine + placebo: Dosing Schedule and Titration of Quetiapine: open-label quetiapine beginning day 1 at 100 mg/day titrated to 400 mg/day by the end of week 1
  Dosing Schedule and Titration of Topiramate:
  All subjects will be randomized to topiramate or matching placebo which will be administered in a double-blind manner.
  Topiramate/Placebo titrated from 25 mg twice daily to 150 mg bid by week 4.
- Quetiapine + Topiramate: Quetiapine + Topiramate
  Quetiapine + Topiramate: Dosing Schedule and Titration of Quetiapine:
  open-label quetiapine beginning day 1 at 100 mg/day titrated to 400 mg/day by the end of week 1
  Dosing Schedule and Titration of Topiramate:
  All subjects will be randomized to topiramate or matching placebo which will be administered in a double-blind manner.
  Topiramate/Placebo titrated from 25 mg twice daily to 150 mg bid by week 4.
Arm/Group | Quetiapine + Placebo | Quetiapine + Topiramate
Number analyzed (Participants) | 21 | 18
Drinks per day | -1.4 (2.3) | -2.4 (5.1)

2. Primary Outcome: Drinks Per Drinking Day
Description: Change in drinks/drinking day (number of drinks consumed divided by the number of days during which alcohol was consumed during that study period)
Time Frame: baseline to 12 weeks or endpoint (up to 11 weeks)
Measure: Mean (Standard Deviation); unit: Drinks per drinking day
Arm/Group | Quetiapine and Placebo | Quetiapine and Topiramate
Number analyzed (Participants) | 21 | 18
Drinks per drinking day | -7.2 (10.2) | -7.3 (6.0)

3. Primary Outcome: Percentage of Days Abstinent
Description: Change in percent days abstinent (the number of non-drinking days divided by the number of days in that study period).
Time Frame: baseline to 12 weeks or endpoint (up to 11 weeks)
Measure: Mean (Standard Deviation); unit: Percentage of days abstinent
Arm/Group | Quetiapine and Placebo | Quetiapine and Topiramate
Number analyzed (Participants) | 21 | 18
Percentage of days abstinent | 15 (19) | 14 (23)

4. Primary Outcome: Percent Heavy Drinking Days
Description: Change in percent heavy drinking days (number of days of > 4 drinks/day divided by number of days in that study period).
Time Frame: baseline to 12 weeks or endpoint (up to 11 weeks)
Measure: Mean (Standard Deviation); unit: Percent heavy drinking days
Arm/Group | Quetiapine and Placebo | Quetiapine and Topiramate
Number analyzed (Participants) | 21 | 18
Percent heavy drinking days | -10 (19) | -14 (25)

ADVERSE EVENTS:
Time Frame: 3 years 9 months
Groups:
- Quetiapine and Placebo: Quetiapine and Placebo
  quetiapine + placebo: Dosing Schedule and Titration of Quetiapine: open-label quetiapine beginning day 1 at 100 mg/day titrated to 400 mg/day by the end of week 1
  Dosing Schedule and Titration of Topiramate:
  All subjects will be randomized to topiramate or matching placebo which will be administered in a double-blind manner.
  Topiramate/Placebo titrated from 25 mg twice daily to 150 mg bid by week 4.
- Quetiapine and Topiramate: Quetiapine and Topiramate
  Quetiapine + Topiramate: Dosing Schedule and Titration of Quetiapine:
  open-label quetiapine beginning day 1 at 100 mg/day titrated to 400 mg/day by the end of week 1
  Dosing Schedule and Titration of Topiramate:
  All subjects will be randomized to topiramate or matching placebo which will be administered in a double-blind manner.
  Topiramate/Placebo titrated from 25 mg twice daily to 150 mg bid by week 4.
Arm/Group | Quetiapine and Placebo | Quetiapine and Topiramate
Serious Adverse Events (participants affected / at risk) | 8/21 | 2/18
Other Adverse Events (participants affected / at risk) | 4/21 | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine and Placebo (N=21) | Quetiapine and Topiramate (N=18)
Suicidal ideation (General disorders) | 7 | 2
Suicide Attempt (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine and Placebo (N=21) | Quetiapine and Topiramate (N=18)
sedation (General disorders) | 4 | 11
Difficulty Arousing (General disorders) | 3 | 9

LIMITATIONS AND CAVEATS:
Additional studies are needed as topiramate has not been systematically assessed. This study was to collect pilot data and more data will need to be collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes